CLINICAL TRIAL: NCT04368078
Title: Lenvatinib Combined Toripalimab in Advanced Hepatocellular Carcinoma: a Single-center, Single-arm, Non-randomized Clinical Study
Brief Title: Lenvatinib Combined Toripalimab in Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-2295
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Toripalimab; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — toripalimab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab plus Lenvatinib (Experimental): Lenvatinib is a novel angiogenesis inhibitor which targets vascular endothelial growth factor 1-3, fibroblast growth factor receptor 1-4, platelet-derived growth factor receptor β, RET and KIT.
  Toripalimab is a recombinant anti-human PD-1 monoclonal antibody.
  Interventions: Drug: Toripalimab plus Lenvatinib

INTERVENTIONS:
Drug: Toripalimab plus Lenvatinib — Toripalimab 240mg, every 3 weeks, intravenous infused, day 1, 6 weeks a cycle. Lenvatinib 8mg (weight<60kg) or 12mg (weight≥60kg), once a day, oral at least 38 days of each 6 weeks cycle, day 2.
  Number of cycle: until progression or unacceptable toxicity events develop
  Other Names: JS001 plus E7080

SUMMARY:
The investigators design a phase IIB clinical study to explore the efficacy and safety of Lenvatinib plus Toripalimab in patients with advanced hepatocellular carcinoma and to analyze potential biomarkers of therapeutic response.

DETAILED DESCRIPTION:
This trial is a single-arm, non-randomized and single-center clinical study of targeted therapy combined immunotherapy in patients with hepatocellular carcinoma.

It is estimated that 76 patients who met the study criteria will be enrolled in Peking Union Medical College Hospital(PUMCH) and treated with Lenvatinib and Toripalimab. The investigators will follow up and collect subjects' data monthly to evaluate the efficacy and safety of treatment, including overall survival and time to progression. Multi-omics data analysis will be used to find potential biomarkers of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Subjects volunteer to participate in the study and agree to sign the informed consent with good compliance and follow-up.
* Subjects are 18 years old or older when signing the informed consent and gender is not limited.
* Imaging (by AASLD or Standard for the diagnosis and treatment of primary liver cancer 2017 in China) or histopathologically or cytologically confirmed advanced Hepatocellular carcinoma.
* BCLC stage B or C. The disease is not suitable for radical surgery and/or topical treatment, or disease progression occurs after surgery and/or local treatment.
* Subjects who have received first-line systemic treatment (targeted therapies other than Lenvatinib, chemotherapy, biological immunotherapy, etc.) except Toripalimab and Lenvatinib could be involved.
* At least one measurable lesion (according to RECIST version 1.1): the measurable lesion has a long diameter ≥ 10 mm or lymphadenpathy has a short diameter ≥ 15 mm in spiral CT scan.
* The ECOG score is 0-1 within 1 week before enrollment.
* Liver function assessment: Child-Pugh Grade A (5-6 points).
* Estimated survival time ≥ 3 months.
* 10. Subjects with HBV infection: HBV DNA<2000 IU/ml or <10^4 copy/mL, and have received anti-HBV therapy for at least 14 days prior to enrollment in the study, subjects with HCV-RNA(+) must receive antiviral therapy;
* Hematology and organ function are sufficient based on the following laboratory results within 14 days prior to the treatment of this study:
* Whole blood cell examination (no blood transfusion within 14 days, no G-CSF use and no drugs use): WBC≥3.0×10^9/L, Hb≥85g/L, ANC≥1.5×10^9/L, PLT≥75×10^9/L.
* Biochemical examination (no ALB infused within 14 days): ALB≥29 g/L, ALP and ALT and AST<5×ULN, TBIL≤3×ULN, creatinine≤1.5×ULN or CCr >50mL/min (standard Cockcroft-Gault formula): Female: CrCl=((140-age) × body weight (kg) × 0.85) / 72 × Serum creatinine (mg/dL); Male: CrCl=((140- age) × body weight (kg) × 1.00) / 72 × Serum creatinine (mg/dL)
* Agree to abstain from sex (avoid heterosexual intercourse) or use contraceptive methods with an annual contraceptive failure rate of less than 1% during treatment and for at least 6 months after the last administration.

Exclusion Criteria:

* Hepatocellular carcinoma patients with any of the following: Suitable for radical surgery; or without an assessment lesion after radical surgery; or liver transplantation history or ready for liver transplantation;
* ECOG score ≥ 2 points.
* Previously received Lenvatinib or Toripalimab treatment.
* History of hepatic encephalopathy.
* Histopathological result show hepatobiliary carcinoma, sarcomatoid liver cancer, mixed cell carcinoma and layered cell carcinoma.
* Already known to be allergic or intolerant to recombinant humanized PD-1 monoclonal antibody drugs (or components) or Lenvatinib.
* Pregnant (positive pregnancy test before taking medicine) or lactating women.
* Received any topical treatment within 4 weeks prior to the study, including but not limited to surgery, radiotherapy, hepatic artery embolization, TACE, hepatic artery perfusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection.
* Previous or existing grade 3 (CTCAE5.0 ) and above gastrointestinal fistula or non-gastrointestinal fistula (such as skin).
* Factors affect Lenvatinib use, such as inability to swallow, chronic diarrhea, intestinal obstruction, or other conditions that significantly affect drug intake and absorption.
* Ascites with clinical symptoms which requires abdominal puncture or drainage therapy, or Child-Pugh score >2.
* Surgery performed within 4 weeks or minor surgery (simple resection or biopsy) within 7 days prior to the trial and patients must be evaluated before the first medication.
* Severe cardiovascular and cerebrovascular diseases, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, cerebrovascular accident or transient ischemic attack, congestive heart failure and arrhythmias within 6 months before enrollment.
* Hepatic and renal dysfunction evidence: jaundice, ascites, and/or bilirubin ≥ 3× ULN, and/or ≥ 3 grade (CTC-AE 5.0) proteinuria (> 3.5g /24 hours), or renal failure requiring blood dialysis or peritoneal dialysis, and / or urine examination shows urinary protein ≥ ++ or 24 hours urine protein >1.0g.
* Persistent >2 grade (CTCAE 5.0) infection.
* Thromboembolism (including stroke and / or transient ischemic attack) within 12 months.
* Hypertension that cannot be controlled well with antihypertensive drugs (systolic blood pressure> 160mmHg, diastolic blood pressure> 100mmHg).
* Already known active central nervous system metastasis and/or cancerous meningitis.
* Active autoimmune disease or autoimmune disease within two years.
* Known central nervous system metastasis and/or cancerous meningitis.
* Prepared or previously received an organ or allogeneic bone marrow transplant
* History of active tuberculosis, such as mycobacterium tuberculosis.
* Gastrointestinal bleeding history in the past 6 months or tendency to gastrointestinal bleeding, such as esophageal varices, local active ulceration lesions, fecal occult blood ≥ (++) (gastroscopy is required when fecal occult blood is (+)).
* History of human immunodeficiency virus infection.
* History of hepatitis B virus or hepatitis C virus infection, and not receive regular treatment.
* Severe non-healing wounds, ulcers or fractures.
* With other malignant tumors within 5 years.
* Previous and current evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonia and severe impairment of lung function.
* Received a potent CYP3A4 inhibitor treatment within 7 days prior to the study or received a potent CYP3A4 inducer within 12 days prior to the study.
* With other active malignant tumor except Hepatocellular carcinoma within 5 years or simultaneously.
* Patients are unsuitable for participation in this research after comprehensive assessment by the researchers.
* Patients participate in another clinical study at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-07-11 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 1 year
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 1 year
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
Progression-free Survival (PFS) | Up to 1 years
  A duration from the date of initial treatment with lenvatinib plus pembrolizumab to disease progression (defined by RECIST 1.1) or death of any cause.
3-months and 6-month Progression free survival rate | Up to 6 months
  Portion of patients who do not experience disease progression (defined by RECIST 1.1) or death of any cause after treated with toripalimab plus lenvatinib for 3 months and 6 months, respectively.
6-months and 1-year mortality rate | Up to 1 years
  Portion of patients who die of any cause after treated with toripalimab plus lenvatinib at 6 months and 1 year, respectively.
Duration of Response (DOR) | Up to 1 years
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Overall Survival (OS) | Up to 2 years
  Duration from the date of initial treatment with lenvatinib plus pembrolizumab to the date of death due to any cause.
clinical benefit rate (CBR) | up to 2 years
  Proportion of patients achieved complete response and partial response for more than 6 months.
Adverse events (AE) | up to 2 years
  Any adverse events related with treatment drugs and details include adverse events type, frequency and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zhao, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Background] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262
- [Background] Llovet JM, Montal R, Villanueva A. Randomized trials and endpoints in advanced HCC: Role of PFS as a surrogate of survival. J Hepatol. 2019 Jun;70(6):1262-1277. doi: 10.1016/j.jhep.2019.01.028. Epub 2019 Mar 31. PMID 30943423
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Boussiotis VA. Molecular and Biochemical Aspects of the PD-1 Checkpoint Pathway. N Engl J Med. 2016 Nov 3;375(18):1767-1778. doi: 10.1056/NEJMra1514296. No abstract available. PMID 27806234
- [Background] Ma W, Gilligan BM, Yuan J, Li T. Current status and perspectives in translational biomarker research for PD-1/PD-L1 immune checkpoint blockade therapy. J Hematol Oncol. 2016 May 27;9(1):47. doi: 10.1186/s13045-016-0277-y. PMID 27234522
- [Background] Jia Y, Zeng Z, Li Y, Li Z, Jin L, Zhang Z, Wang L, Wang FS. Impaired function of CD4+ T follicular helper (Tfh) cells associated with hepatocellular carcinoma progression. PLoS One. 2015 Feb 17;10(2):e0117458. doi: 10.1371/journal.pone.0117458. eCollection 2015. PMID 25689070
- [Background] Finn RS, Ryoo BY, Merle P, Kudo M, Bouattour M, Lim HY, Breder V, Edeline J, Chao Y, Ogasawara S, Yau T, Garrido M, Chan SL, Knox J, Daniele B, Ebbinghaus SW, Chen E, Siegel AB, Zhu AX, Cheng AL; KEYNOTE-240 investigators. Pembrolizumab As Second-Line Therapy in Patients With Advanced Hepatocellular Carcinoma in KEYNOTE-240: A Randomized, Double-Blind, Phase III Trial. J Clin Oncol. 2020 Jan 20;38(3):193-202. doi: 10.1200/JCO.19.01307. Epub 2019 Dec 2. PMID 31790344
- [Background] Gunda V, Gigliotti B, Ashry T, Ndishabandi D, McCarthy M, Zhou Z, Amin S, Lee KE, Stork T, Wirth L, Freeman GJ, Alessandrini A, Parangi S. Anti-PD-1/PD-L1 therapy augments lenvatinib's efficacy by favorably altering the immune microenvironment of murine anaplastic thyroid cancer. Int J Cancer. 2019 May 1;144(9):2266-2278. doi: 10.1002/ijc.32041. Epub 2019 Jan 24. PMID 30515783
- [Background] Kato Y, Tabata K, Kimura T, Yachie-Kinoshita A, Ozawa Y, Yamada K, Ito J, Tachino S, Hori Y, Matsuki M, Matsuoka Y, Ghosh S, Kitano H, Nomoto K, Matsui J, Funahashi Y. Lenvatinib plus anti-PD-1 antibody combination treatment activates CD8+ T cells through reduction of tumor-associated macrophage and activation of the interferon pathway. PLoS One. 2019 Feb 27;14(2):e0212513. doi: 10.1371/journal.pone.0212513. eCollection 2019. PMID 30811474
- [Background] Makker V, Rasco D, Vogelzang NJ, Brose MS, Cohn AL, Mier J, Di Simone C, Hyman DM, Stepan DE, Dutcus CE, Schmidt EV, Guo M, Sachdev P, Shumaker R, Aghajanian C, Taylor M. Lenvatinib plus pembrolizumab in patients with advanced endometrial cancer: an interim analysis of a multicentre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2019 May;20(5):711-718. doi: 10.1016/S1470-2045(19)30020-8. Epub 2019 Mar 25. PMID 30922731
- [Background] Tang B, Yan X, Sheng X, Si L, Cui C, Kong Y, Mao L, Lian B, Bai X, Wang X, Li S, Zhou L, Yu J, Dai J, Wang K, Hu J, Dong L, Song H, Wu H, Feng H, Yao S, Chi Z, Guo J. Safety and clinical activity with an anti-PD-1 antibody JS001 in advanced melanoma or urologic cancer patients. J Hematol Oncol. 2019 Jan 14;12(1):7. doi: 10.1186/s13045-018-0693-2. PMID 30642373
- [Background] Sheng X, Yan X, Chi Z, Si L, Cui C, Tang B, Li S, Mao L, Lian B, Wang X, Bai X, Zhou L, Kong Y, Dai J, Wang K, Tang X, Zhou H, Wu H, Feng H, Yao S, Flaherty KT, Guo J. Axitinib in Combination With Toripalimab, a Humanized Immunoglobulin G4 Monoclonal Antibody Against Programmed Cell Death-1, in Patients With Metastatic Mucosal Melanoma: An Open-Label Phase IB Trial. J Clin Oncol. 2019 Nov 10;37(32):2987-2999. doi: 10.1200/JCO.19.00210. Epub 2019 Aug 12. PMID 31403867
- [Background] Hodi FS, Ballinger M, Lyons B, Soria JC, Nishino M, Tabernero J, Powles T, Smith D, Hoos A, McKenna C, Beyer U, Rhee I, Fine G, Winslow N, Chen DS, Wolchok JD. Immune-Modified Response Evaluation Criteria In Solid Tumors (imRECIST): Refining Guidelines to Assess the Clinical Benefit of Cancer Immunotherapy. J Clin Oncol. 2018 Mar 20;36(9):850-858. doi: 10.1200/JCO.2017.75.1644. Epub 2018 Jan 17. PMID 29341833